CLINICAL TRIAL: NCT07332871
Title: Safety and efficacY of conductioN System paCing and Atrioventricular Junctional Ablation Combined With ICD Implantation in Patients With End-stage Heart Failure and Atrial Fibrillation Eligible for Heart Transplantation (SYNC AF-HTx) : Multicenter Prospective Randomized Controlled Trial
Brief Title: Conduction System Pacing and AV Junction Ablation in Heart Failure With Atrial Fibrillation (SYNC AF-HTx)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2025-1357
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Atrial Fibrillation; Defibrillators, Implantable
Keywords: Left Bundle Branch Pacing (LBBP); Conduction System Pacing (CSP); Atrioventricular Junction Ablation (AVJ ablation); End-stage Heart Failure; Heart Transplantation; ICD
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYNC group (Experimental): Combined procedure of ICD implantation, LBBP lead insertion, and AVJ ablation.
  Interventions: Device: LBBP + AVJ Ablation with ICD
- Control group (Active Comparator): Standard ICD implantation with minimal ventricular pacing strategy.
  Interventions: Device: ICD Only

INTERVENTIONS:
Device: LBBP + AVJ Ablation with ICD — Insertion of an LBBP lead (Medtronic SelectSecure™ 3830) and performing AVJ ablation to ensure heart rate regularization and ventricular synchronization
  Arms: SYNC group
Device: ICD Only — Participants receive standard ICD implantation with a minimal ventricular pacing strategy
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of conduction system pacing (CSP) using left bundle branch pacing (LBBP) and atrioventricular junction (AVJ) ablation in patients with end-stage heart failure and permanent atrial fibrillation (AF). Participants who are candidates for heart transplantation or left ventricular assist device (LVAD) implantation will be randomized to either the SYNC group (ICD implantation combined with LBBP and AVJ ablation) or the control group (ICD implantation only). The investigators will compare clinical outcomes, including mortality and heart failure hospitalization, between the two strategies over a 1-year follow-up period.

DETAILED DESCRIPTION:
End-stage heart failure patients often face a poor prognosis due to comorbid permanent AF, which leads to irregular heart rates and worsens ventricular function. While implantable cardioverter-defibrillators (ICDs) are standard for preventing sudden cardiac death, they may not sufficiently prevent heart failure progression in patients with narrow QRS complexes. This study explores a "SYNC" strategy using LBBP and AVJ ablation to achieve ventricular synchronization and heart rate regularization. This is a multicenter, prospective, randomized (1:1), single-blind trial involving 120 participants.

Inclusion Criteria: Participants must have LVEF≤35%, permanent AF for >6 months, and be eligible for ICD implantation while awaiting heart transplantation or LVAD.

Intervention (SYNC Group): Participants receive an ICD with an LBBP lead (Medtronic SelectSecure™ 3830) and undergo AVJ ablation.

Control Group: Participants receive standard ICD implantation with a minimal ventricular pacing setting.

Follow-up: Clinical assessments, echocardiography, and device profiles will be monitored at baseline, 1, 3, 6, and 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

Candidates for ICD implantation (primary or secondary prevention). Permanent AF (>6 months) unsuitable for or failed catheter ablation. End-stage heart failure considering heart transplant or LVAD. LVEF ≤ 35 within 6 weeks before enrollment. NYHA functional class ≥ II. On GDMT for at least 3 months. Age ≥ 19 years.

Exclusion Criteria:

Existing LVAD or prior heart transplantation. Indications for cardiac resynchronization therapy (CRT). History of mechanical tricuspid valve replacement. Expected survival≤ 12 months. Inability to comply with the study protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality, heart failure hospitalization, or urgent heart transplantation | Time Frame: Up to 12 months
  Occurrence of the first event among the composite components

SECONDARY OUTCOMES:
All cause mortality | Up to 12 months
  All cause deaths including cardiovascular and non-cardiovascular deaths.
Cardiovascular mortality | Up to 12 months
  Cardiovascular death
Heart failure hospitalization | Up to 12 months
  An unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required intravenous therapy.
Urgent heart transplantation | Up to 12 months
  Urgent heart transplantation
LV systolic function | 6months and 12months
  LVEF measure by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei University College of Medicine., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided